CLINICAL TRIAL: NCT05863507
Title: The Influence of Daily Grapes Intake on Sarcopenia in Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: California Table Grape Commission (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1867416
Record Dates: First submitted 2023-04-26; First posted 2023-05-18 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Sarcopenia
MeSH Terms: conditions — Sarcopenia

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- grape group (Experimental): The participant of this group will received a lyophilized grape powder
  Interventions: Dietary Supplement: Grape powder supplementation
- placebo group (Placebo Comparator): The participant of this group will received a lyophilized powder similar to the grape one
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Grape powder supplementation — The participants will be willing to consume the grape powder dissolve in water daily for 6 weeks
  Arms: grape group
Dietary Supplement: Placebo — The participants will be willing to consume the placebo powder, similar to the grape powder, dissolve in water daily for 6 weeks
  Arms: placebo group

SUMMARY:
Sarcopenia, characterized by loss of muscle mass and function, is a prevalent disorder in elderly individuals or individuals with chronic diseases. Given the above, there is an ongoing intensive search for novel therapies, including dietary ones, that can attenuate the loss of muscle mass and strength in the elderly. A proposed mechanism by which skeletal muscles might mediate their protective effect against sarcopenia is by secreting myokines as irisin. Phenolic compounds presents in grape have shown to be able to induce irisin secretion in muscle from rats supplemented with a grape pomace extract. The Ian of this study is to evaluate this mechanism in humans.

DETAILED DESCRIPTION:
Scientific rationale Sarcopenia, characterized by loss of muscle mass and function, is a prevalent disorder in elderly individuals or individuals with chronic diseases. It leads to fragility and disability, worsens the prognosis of many diseases, and significantly enhances morbidity and mortality. With the increasing life expectancy and rapid growth of the aged population, sarcopenia is becoming an emerging public health issue with huge socioeconomic burden.

Given the above, there is an ongoing intensive search for novel therapies, including dietary ones, that can attenuate the loss of muscle mass and strength in the elderly. Interestingly, a growing body of research indicate that nutritional factors can preserve muscle function from age- related decline. In particular, phenolic compounds, widely distributed in fruits including grapes, have shown beneficial effects in muscle health. However, the exact influence of grapes and grapes phenolic compounds mitigating sarcopenia in humans remains unexplored.

A proposed mechanism by which skeletal muscles might mediate their protective effect against sarcopenia is by secreting myokines. Irisin is a myokine regulated by peroxisome proliferator- activated receptor gamma co-activator-1α (PGC-1α) and released into the bloodstream after cleavage of the Fibronectin type III domain-containing protein 5 (FNDC5). Recent studies have indicated that circulating irisin can promote skeletal muscle growth. Lower irisin concentrations have been observed in sarcopenia patients and dialyzed patients with cardiovascular disease. Furthermore, lower irisin plasma levels are associated with sarcopenia in postmenopausal women.

In a recent study, it have been shown that phenolic compounds present in a grape pomace extract (GPE), rich in phenolic compounds, prevent irisin downregulation in rats fed a high-fat diet and in L6 myotube cells. In particular, we documented that consumption of the GPE activates the FNDC5/irisin pathway, increased AMPK phosphorylation in skeletal muscle and increased irisin plasma levels. These data strongly indicate that phenolic compounds enhance irisin levels in vitro and in vivo. These intriguing data allow us to hypothesize that phenolic compounds present in grapes might prevent sarcopenia in elderly humans, in part, by increasing irisin levels.

Specific objectives

The objective of this proposal is to evaluate whether the daily consumption of a freeze-dried table grape powder, rich in phenolic compounds, mitigates sarcopenia in postmenopausal women. The hypothesis is that daily dietary supplementation with a grape powder improves health span, mitigates sarcopenia parameters and increases irisin plasma levels in postmenopausal women. To test this hypothesis, the following aims will be pursued:

* To determine the efficacy of a freeze-dried table grape powder, rich in phenolic compounds, to mitigate sarcopenia parameters in postmenopausal women.
* To evaluate the effect of a freeze-dried table grape powder on key metabolic regulators of sarcopenia in postmenopausal women.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women aged 60 years and older
* Normal BMI with values between 18.4 and 24.9 kg/m2
* Hand-grip strength media value of 16 kg or lower
* Blood pressure below 130/80 mmHg, and plasma glucose and cholesterol concentrations below 100 and 200 mg/dl.

Exclusion Criteria:

* History of specific muscle diseases
* Peripheral vascular disease
* Intermittent claudication
* Central and peripheral nervous system disorders
* Cachexia
* Active diagnosis of diabetes mellitus
* Myocardial infarction
* Stroke
* Liver disease
* Dialysis
* Long-term steroid therapy
* Actively receiving treatment for cancer or severe infection (excluding short-term antibiotic therapy)
* Weight less than 140 pounds
* Anemia and blood donations in the past 30 days.
* Participants should not be taking dietary supplements at the time of the study

Min Age: 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 15 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2024-07-14 (Actual); Study Completion 2024-07-14 (Actual)

PRIMARY OUTCOMES:
Plasma irisin levels | 6 weeks
  The investigators will measure irisin levels in plasma

CONTACTS AND LOCATIONS:
Overall Officials: Francene G Steinberg, PhD, Study Chair — University of California, Davis
Locations (1):
- Nutrition Department, Ragle Facility University of California, Davis, Davis, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2022-08-25): https://cdn.clinicaltrials.gov/large-docs/07/NCT05863507/Prot_ICF_000.pdf